CLINICAL TRIAL: NCT03151343
Title: Effects of SGLT-2 Inhibitor on Myocardial Perfusion, Function and Metabolism in Type 2 DM Patients at High Cardiovascular Risk: The SIMPle Randomized Clinical Trial
Brief Title: SGLT-2 Inhibitor and Myocardial Perfusion, Function and Metabolism in T2 DM Patients at High Cardiovascular Risk
Acronym: SIMPLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Caroline M Kistorp (Other)
Collaborators: Danish Heart Foundation (Other); Herlev and Gentofte Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Caroline M Kistorp, Principal Investigator, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-775; 2016-003743-10 (EudraCT Number)
Record Dates: First submitted 2017-03-12; First posted 2017-05-12 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Participants will be treated with either empagliflozin or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Experimental): Empagliflozin, coated tablets, 25mg, once daily, for 13 weeks
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Placebo, coated tablets, once daily, for 13 weeks
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin tablet
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo Oral Tablet — Sugar pill, visually identical to active comparator
  Arms: Placebo

SUMMARY:
Patients with type 2 diabetes (T2 DM) have a markedly increased risk of heart disease and it is estimated that, in the danish population, up 80% percent of patients with type 2 diabetes die from heart disease.

The sodium glucose cotransport-2 (SGLT-2) inhibitors were developed as an anti-diabetic therapy reducing blood glucose and weight by decreasing glucose reabsorption in the kidneys, leading to glucose excretion via the urine. However, in 2015 the EMPA-REG study showed that treatment with the SGLT-2 inhibitor empagliflozin significantly reduced the cardiovascular mortality and risk of admission under the diagnosis of heart failure in a population of patients with type 2 diabetes in addition to other risk factors for heart disease. The mechanism behind this surprising result is unknown and warrants further study.

The primary hypothesis of the present study is that treatment with empagliflozin improves the function and blood supply of the heart muscle cells in patients with type 2 diabetes and high risk of heart disease. The investigators will test this hypothesis by enrolling 92 participants with type 2 diabetes and other risk factors for heart disease, and treating them with either empagliflozin or a placebo. During the study period the investigators will monitor the effects of the treatment with various techniques such as heart scans using CT and ultrasound, measurements of the fluid pressures in the heart chambers, body composition measurements and a variety of relevant blood test.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of type 2 diabetes mellitus at least 3 months prior to baseline visit
* For patients on background therapy: stable dose of anti-diabetics within 30 days prior to baseline
* HbA1c of ≥6.5% and ≤10% at screening for patients on background therapy or HbA1c of ≥6.5 % and ≤ 9.0% at screening for drug-naïve patients.
* BMI ≤ 45 kg/m2 at screening
* Age ≥18 years
* Negative pregnancy test (fertile women). Fertile women must use safe contraceptives (spiral, hormonal contraceptives) for the duration of the study
* Able to understand the written patient information and to give informed consent
* Patients must have high cardiovascular risk, defined as at least one of the following:
* Albuminuria ( albumin/creatinine ratio ≥ 30 mg/g or plasma NT-proBNP ≥ 70 pg/ml)
* Confirmed history of myocardial infarction (>2 months prior to baseline)
* Heart failure according to the Framingham Heart Failure Criteria
* Or patient discharged from hospital with a documented diagnosis of unstable angina within 12 months prior to baseline
* Evidence of coronary artery disease by CAG in 1 or more major coronary arteries

OR at least one of the following: a positive noninvasive stress test, or A positive stress echocardiography showing regional systolic wall motion abnormalities, or A positive scintigraphic test showing stress-induced ischemia,

* History of ischemic or haemorrhagic stroke (>2 months prior to informed consent)
* Presence of peripheral artery disease (symptomatic or not ) documented by either: previous limb angioplasty, stenting or bypass surgery; or previous limb or foot amputation due to circulatory insufficiency; or angiographic evidence of significant (> 50%) peripheral artery stenosis in at least one limb; or evidence from a non-invasive measurement of significant (>50% or as reported as hemodynamically significant) peripheral artery stenosis in at least one limb; or ankle brachial index of < 0.9

Exclusion Criteria:

* Allergic to the study medication
* Treatment with SGLT-2 inhibitor within 3 months prior to baseline
* Impaired kidney function, eGFR ≤ 30 ml/min
* Severe liver insufficiency (Child-Pugh class C)
* ECG showing malign ventricular arrhythmia or prolonged QT-interval (>500ms)
* Untreated clinical significant heart valve disease
* Planned cardiac surgery or angioplasty within 3 months.
* Myocardial infarction (MI) ≤ 30 days prior to baseline
* Percutaneous coronary intervention (PCI) ≤ 4 weeks prior to baseline
* History of coronary artery bypass graft (CABG) ≤ 8 weeks prior to enrollment
* Prior history of heart transplantation
* Unstable angina, known severe left main coronary artery stenosis, severe heart failure, uncontrolled arrhythmias, symptomatic hypotension or severe hypertension (systolic blood pressure < 90 or > 180 mmHg, respectively), sick sinus syndrome or > 1st degree atrioventricular block in the absence of a functioning pacemaker
* Requirement of emergent cardiac medical intervention or catheterization
* Treatment with theophylline, or theophylline containing medications
* History of known or suspected bronchoconstrictive or bronchospastic lung disease (e.g., asthma)
* Pregnancy or desire hereof or breastfeeding.

Additional exclusion criteria for hemodynamics substudy

* LVEF ≤ 40 % evaluated at baseline echocardiography
* Inability to perform a VO2 max test
* Hypertrophic cardiomyopathy
* Left ventricular assist device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Rb-82 PET | 13 weeks
  Between group difference in the change in myocardial flow reserve (MFR) by Rb-82 PET. Measured as change in global perfusion from rest to adenosine-induced stress.
Invasive hemodynamics | 13 weeks
  Substudy, performed on 38 participants from the main group. Using right heart catheterisation to measure between group difference in the change in pulmonary capillary weight pressure (PCWP) at 25 watts (supine bicycle ergometer)

SECONDARY OUTCOMES:
Echocardiography | 13 weeks
  Between group difference in the change in global left ventricular function assessed by echocardiography
GFR | 13 weeks
  Between group difference in the change in renal function assessed by Cr-51 EDTA
U-alb/crea | 13 weeks
  Between group difference in the change urinary albumin/creatinine ratio
24 hour BP | 13 weeks
  Between group difference in the change in 24 hour BP
Pulse wave analysis | 13 weeks
  Between group difference in the change in pulse wave analysis
Insulin resistance | 13 weeks
  Between group difference in the changes in insulin resistance by Matsuda index
Insulin resistance | 13 weeks
  Between group difference in the changes in insulin resistance by HOMA
Biomarkers | 13 weeks
  Between group difference in the change in NT-proBNP, MR-proANP, MR-proADM, GAL-3, hsTNT, GDF-15, PIGF, sFlt-1, FFA, ADPN, leptin, TNF-α, IL-6, MCP-1, MAC-1, COLL-A1, FGF-21, beta-hydroxybutyrate, AGEs CML, sRAGE
Questionnaires | 13 weeks
  Between group difference in the change in Health status, assessed by the EuroQol EQ-5D-5L questionnaire
Questionnaires, continued | 13 weeks
  Between group difference in the change in Health status, assessed by the Minnesota Living with Heart Failure questionnaire
DEXA | 13 weeks
  Between group difference in the change in body composition by DEXA scan
Invasive hemodynamics - continued | 13 weeks
  Between group difference in the change in CO at rest, 25 watts and peak exercise
Invasive hemodynamics - continued | 13 weeks
  Between group difference in the change in CVP at rest, 25 watts and peak exercise
Invasive hemodynamics - continued | 13 weeks
  Between group difference in the change in PCWP at rest, 25 watts and peak exercise
Invasive hemodynamics - continued | 13 weeks
  Between group difference in the change in PAP at rest, 25 watts and peak exercise
Invasive hemodynamics - continued | 13 weeks
  Between group difference in the change in SvO2 at rest, 25 watts and peak exercise
Adipose tissue | 13 weeks
  Between group difference in the changes in levels of adipocyte differentiation
Adipose tissue | 13 weeks
  Between group difference in the changes in macrophage infiltration
Adipose tissue | 13 weeks
  Between group difference in the changes in extracellular matrix fibrosis
Daily activity | 13 weeks
  Between group difference in the change in daily activity levels measured by patient-worn accelerometers.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M Kistorp, MD, PhD., Principal Investigator — Herlev og Gentofte Hospital
Locations (1):
- Herlev og Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No
Any sharing of data must be approved by the regional ethics committee, and at the time of protocol writing there was no justification for data sharing outside of the current project

REFERENCES:
- [Background] Gallo LA, Wright EM, Vallon V. Probing SGLT2 as a therapeutic target for diabetes: basic physiology and consequences. Diab Vasc Dis Res. 2015 Mar;12(2):78-89. doi: 10.1177/1479164114561992. Epub 2015 Jan 23. PMID 25616707
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Lin B, Koibuchi N, Hasegawa Y, Sueta D, Toyama K, Uekawa K, Ma M, Nakagawa T, Kusaka H, Kim-Mitsuyama S. Glycemic control with empagliflozin, a novel selective SGLT2 inhibitor, ameliorates cardiovascular injury and cognitive dysfunction in obese and type 2 diabetic mice. Cardiovasc Diabetol. 2014 Oct 26;13:148. doi: 10.1186/s12933-014-0148-1. PMID 25344694
- [Background] deKemp RA, Yoshinaga K, Beanlands RS. Will 3-dimensional PET-CT enable the routine quantification of myocardial blood flow? J Nucl Cardiol. 2007 May-Jun;14(3):380-97. doi: 10.1016/j.nuclcard.2007.04.006. PMID 17556173
- [Background] Naya M, Murthy VL, Foster CR, Gaber M, Klein J, Hainer J, Dorbala S, Blankstein R, Di Carli MF. Prognostic interplay of coronary artery calcification and underlying vascular dysfunction in patients with suspected coronary artery disease. J Am Coll Cardiol. 2013 May 21;61(20):2098-106. doi: 10.1016/j.jacc.2013.02.029. Epub 2013 Mar 21. PMID 23524053
- [Background] Dorbala S, Di Carli MF, Beanlands RS, Merhige ME, Williams BA, Veledar E, Chow BJ, Min JK, Pencina MJ, Berman DS, Shaw LJ. Prognostic value of stress myocardial perfusion positron emission tomography: results from a multicenter observational registry. J Am Coll Cardiol. 2013 Jan 15;61(2):176-84. doi: 10.1016/j.jacc.2012.09.043. Epub 2012 Dec 5. PMID 23219297
- [Background] Sattar N, McLaren J, Kristensen SL, Preiss D, McMurray JJ. SGLT2 Inhibition and cardiovascular events: why did EMPA-REG Outcomes surprise and what were the likely mechanisms? Diabetologia. 2016 Jul;59(7):1333-1339. doi: 10.1007/s00125-016-3956-x. Epub 2016 Apr 25. PMID 27112340
- [Background] Hasenfuss G, Hayward C, Burkhoff D, Silvestry FE, McKenzie S, Gustafsson F, Malek F, Van der Heyden J, Lang I, Petrie MC, Cleland JG, Leon M, Kaye DM; REDUCE LAP-HF study investigators. A transcatheter intracardiac shunt device for heart failure with preserved ejection fraction (REDUCE LAP-HF): a multicentre, open-label, single-arm, phase 1 trial. Lancet. 2016 Mar 26;387(10025):1298-304. doi: 10.1016/S0140-6736(16)00704-2. PMID 27025436
- [Background] Ersboll M, Valeur N, Mogensen UM, Andersen M, Greibe R, Moller JE, Hassager C, Sogaard P, Kober L. Global left ventricular longitudinal strain is closely associated with increased neurohormonal activation after acute myocardial infarction in patients with both reduced and preserved ejection fraction: a two-dimensional speckle tracking study. Eur J Heart Fail. 2012 Oct;14(10):1121-9. doi: 10.1093/eurjhf/hfs107. Epub 2012 Jun 28. PMID 22753861
- [Background] Jhund PS, Anand IS, Komajda M, Claggett BL, McKelvie RS, Zile MR, Carson PE, McMurray JJ. Changes in N-terminal pro-B-type natriuretic peptide levels and outcomes in heart failure with preserved ejection fraction: an analysis of the I-Preserve study. Eur J Heart Fail. 2015 Aug;17(8):809-17. doi: 10.1002/ejhf.274. Epub 2015 Apr 29. PMID 25921853
- [Background] Sharma S, Adrogue JV, Golfman L, Uray I, Lemm J, Youker K, Noon GP, Frazier OH, Taegtmeyer H. Intramyocardial lipid accumulation in the failing human heart resembles the lipotoxic rat heart. FASEB J. 2004 Nov;18(14):1692-700. doi: 10.1096/fj.04-2263com. PMID 15522914
- [Background] Ferrannini E, Muscelli E, Frascerra S, Baldi S, Mari A, Heise T, Broedl UC, Woerle HJ. Metabolic response to sodium-glucose cotransporter 2 inhibition in type 2 diabetic patients. J Clin Invest. 2014 Feb;124(2):499-508. doi: 10.1172/JCI72227. Epub 2014 Jan 27. PMID 24463454
- [Background] Ferrannini E, Baldi S, Frascerra S, Astiarraga B, Heise T, Bizzotto R, Mari A, Pieber TR, Muscelli E. Shift to Fatty Substrate Utilization in Response to Sodium-Glucose Cotransporter 2 Inhibition in Subjects Without Diabetes and Patients With Type 2 Diabetes. Diabetes. 2016 May;65(5):1190-5. doi: 10.2337/db15-1356. Epub 2016 Feb 9. PMID 26861783
- [Background] Mudaliar S, Alloju S, Henry RR. Can a Shift in Fuel Energetics Explain the Beneficial Cardiorenal Outcomes in the EMPA-REG OUTCOME Study? A Unifying Hypothesis. Diabetes Care. 2016 Jul;39(7):1115-22. doi: 10.2337/dc16-0542. PMID 27289124
- [Background] Ferrannini E, Mark M, Mayoux E. CV Protection in the EMPA-REG OUTCOME Trial: A "Thrifty Substrate" Hypothesis. Diabetes Care. 2016 Jul;39(7):1108-14. doi: 10.2337/dc16-0330. PMID 27289126
- [Background] Aubert CE, Michel PL, Gillery P, Jaisson S, Fonfrede M, Morel F, Hartemann A, Bourron O. Association of peripheral neuropathy with circulating advanced glycation end products, soluble receptor for advanced glycation end products and other risk factors in patients with type 2 diabetes. Diabetes Metab Res Rev. 2014 Nov;30(8):679-85. doi: 10.1002/dmrr.2529. PMID 24449227
- [Background] Willemsen S, Hartog JW, van Veldhuisen DJ, van der Meer P, Roze JF, Jaarsma T, Schalkwijk C, van der Horst IC, Hillege HL, Voors AA. The role of advanced glycation end-products and their receptor on outcome in heart failure patients with preserved and reduced ejection fraction. Am Heart J. 2012 Nov;164(5):742-749.e3. doi: 10.1016/j.ahj.2012.07.027. PMID 23137505
- [Background] Hartog JW, Voors AA, Bakker SJ, Smit AJ, van Veldhuisen DJ. Advanced glycation end-products (AGEs) and heart failure: pathophysiology and clinical implications. Eur J Heart Fail. 2007 Dec;9(12):1146-55. doi: 10.1016/j.ejheart.2007.09.009. PMID 18023248
- [Background] Oelze M, Kroller-Schon S, Welschof P, Jansen T, Hausding M, Mikhed Y, Stamm P, Mader M, Zinssius E, Agdauletova S, Gottschlich A, Steven S, Schulz E, Bottari SP, Mayoux E, Munzel T, Daiber A. The sodium-glucose co-transporter 2 inhibitor empagliflozin improves diabetes-induced vascular dysfunction in the streptozotocin diabetes rat model by interfering with oxidative stress and glucotoxicity. PLoS One. 2014 Nov 17;9(11):e112394. doi: 10.1371/journal.pone.0112394. eCollection 2014. PMID 25402275
- [Background] Jorgensen RM, Levitan J, Halevi Z, Puzanov N, Abildstrom SZ, Messier MD, Huikuri HV, Haarbo J, Thomsen PE, Jons C; CARISMA investigators. Heart rate variability density analysis (Dyx) for identification of appropriate implantable cardioverter defibrillator recipients among elderly patients with acute myocardial infarction and left ventricular systolic dysfunction. Europace. 2015 Dec;17(12):1848-54. doi: 10.1093/europace/euu394. Epub 2015 Mar 8. PMID 25755288
- [Background] Ruwald AC, Bloch Thomsen PE, Gang U, Jorgensen RM, Huikuri HV, Jons C. New-onset atrial fibrillation predicts malignant arrhythmias in post-myocardial infarction patients--a Cardiac Arrhythmias and RIsk Stratification after acute Myocardial infarction (CARISMA) substudy. Am Heart J. 2013 Nov;166(5):855-63.e3. doi: 10.1016/j.ahj.2013.08.017. Epub 2013 Sep 26. PMID 24176441
- [Background] Ridderstrale M, Andersen KR, Zeller C, Kim G, Woerle HJ, Broedl UC; EMPA-REG H2H-SU trial investigators. Comparison of empagliflozin and glimepiride as add-on to metformin in patients with type 2 diabetes: a 104-week randomised, active-controlled, double-blind, phase 3 trial. Lancet Diabetes Endocrinol. 2014 Sep;2(9):691-700. doi: 10.1016/S2213-8587(14)70120-2. Epub 2014 Jun 16. PMID 24948511
- [Background] von Scholten BJ, Hasbak P, Christensen TE, Ghotbi AA, Kjaer A, Rossing P, Hansen TW. Cardiac (82)Rb PET/CT for fast and non-invasive assessment of microvascular function and structure in asymptomatic patients with type 2 diabetes. Diabetologia. 2016 Feb;59(2):371-8. doi: 10.1007/s00125-015-3799-x. Epub 2015 Nov 2. PMID 26526662
- [Derived] Wolsk E, Jurgens M, Schou M, Ersboll M, Hasbak P, Kjaer A, Zerahn B, Brandt NH, Gaede PH, Rossing P, Faber J, Inzucchi SE, Kistorp CM, Gustafsson F. Randomized Controlled Trial of the Hemodynamic Effects of Empagliflozin in Patients With Type 2 Diabetes at High Cardiovascular Risk: The SIMPLE Trial. Diabetes. 2022 Apr 1;71(4):812-820. doi: 10.2337/db21-0721. PMID 35061894
- [Derived] Jurgens M, Schou M, Hasbak P, Kjaer A, Wolsk E, Zerahn B, Wiberg M, Brandt NH, Gaede PH, Rossing P, Faber J, Inzucchi S, Gustafsson F, Kistorp CM. Design of a randomised controlled trial of the effects of empagliflozin on myocardial perfusion, function and metabolism in type 2 diabetes patients at high cardiovascular risk (the SIMPLE trial). BMJ Open. 2019 Nov 27;9(11):e029098. doi: 10.1136/bmjopen-2019-029098. PMID 31780586